CLINICAL TRIAL: NCT05520398
Title: Cognitive and Neural Networks in Psychiatry (CNNP): Neural Mechanisms of Obsessive-compulsive Disorder (OCD) Treatment Failure (ERP in Silico)
Brief Title: Neural Mechanisms of Obsessive-compulsive Disorder (OCD) Treatment Failure
Acronym: ERP in Silico
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0541
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to understand why patients with obsessive-compulsive disorder (OCD) fail in therapy.

To understand the neural mechanisms involved in exposure therapy that support success and clinical improvement in order to improve therapy outcomes for OCD patients.

DETAILED DESCRIPTION:
A course of therapy is recommended for individuals with obsessive-compulsive disorder (OCD). It is usually a type of cognitive behavioural therapy (CBT) with exposure and response prevention (ERP).

In this study the investigators assess patients pre-therapy and post-therapy evaluating symptom severity (measured by the Y-BOCS) and decision-making (measured by online questionnaires and computer-based behavioural tasks).

To examine how decisions are formed in patients undergoing OCD CBT, how behaviour changes after a non-pharmacological therapy module and how it is associated to the alleviation of OCD symptoms.

The study, which will recruit 90 patients, is based at University College London - Wellcome Centre for Human Neuroimaging. This study is a part of the Cognitive and Neural Networks in Psychiatry (CNNP) study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obsessive-compulsive disorder (OCD)
* Fluent in written and spoken English
* Normal/corrected to normal vision
* Expecting to start OCD therapy

Exclusion Criteria:

* Autism spectrum disorder, psychosis, schizophrenia, addiction, substance abuse, bipolar, hoarding, or Tourette disorder
* Hearing conditions: tinnitus, ear inflammation, hearing sensitivity, hearing loss, requires hearing aids
* Colour blindness
* Severe learning disabilities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with obsessive-compulsive disorder (OCD)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown obsessive compulsive scale (Y-BOCS) | 3 - 9 months
  The Y-BOCS is a 10-item scale used to assess symptom severity in OCD.
Decision making and learning tasks | 3 - 9 months
  Computer-based behavioural task developed by the investigators to understand decision making in OCD.

SECONDARY OUTCOMES:
Patient EX/RP Adherence Scale (PEAS) | 3 - 9 months
  Self-report assessment for patient's therapy adherence.
Short form of Obsessive Beliefs Questionnaire (OBQ) | 3 - 9 months
  Self-report assessment for obsessive beliefs.
Brief Experiential Avoidance Questionnaire (BEAQ) | 3 - 9 months
  Self-report assessment for experiential avoidance.
International Cognitive Ability Resource (ICAR16) | 3 - 9 months
  Measure to assess cognitive ability.
Worry Domains Questionnaire - Short Form (WDQ-SF) | 3 - 9 months
  Self-report assessment for worry.
The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | 3 - 9 months
  Self-report assessment for quality of life assessment.
Sheehan Disability Scale (SDS) | 3 - 9 months
  Self-report assessment for functional impairment.
State-Trait Anxiety Inventory (STAI) | 3 - 9 months
  Measure of trait and state anxiety
Zung Self-Rating Depression Scale (SDS) | 3 - 9 months
  Self-report measure of depressive symptomatology.
Anxiety Sensitivity Index (ASI-3) | 3 - 9 months
  Self-report measure for anxiety sensitivity symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hauser, PhD, Principal Investigator — University College, London
Locations (1):
- Max Planck UCL Centre for Computational Psychiatry and Ageing Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided